CLINICAL TRIAL: NCT06232889
Title: Deuterium Metabolic MRI and [18F]-Flourodesoxyglucose Positron Emission Tomography for Assessment of Treatment Response Following Radioembolization; Pilot Study
Brief Title: Deuterium Metabolic MRI and [18F]FDG PET for Assessment of Treatment Response Following Radioembolization
Acronym: DEPLETE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Arthur Braat, Dr. A.J.A.T. Braat, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DEPLETE
Record Dates: First submitted 2024-01-12; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Fluorodeoxyglucose F18; Phosphoric Monoester Hydrolases; Phosphoric Diester Hydrolases
Keywords: FDG-PET; 31P spectroscopy; MRI; Deuterium Metabolic Imaging; SIRT; TARE; Radioembolization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Deuterium Glucose Metabolic Imaging with MRI spectroscopy — MRI spectroscopy of the liver, following ingestion of 20 mg deuterium glucose p.o., prior to and after radioembolization treatment for mCRC

SUMMARY:
Radioembolization, also known as Selective Internal Radiation Therapy (SIRT), is a liver-directed therapy for patients suffering from hepatic metastases. As SIRT is a liver-directed treatment, only patients with liver-only or liver-dominant disease are eligible for treatment. FDG-PET/CT is known to outperform conventional anatomical imaging modalities (CT or MRI) for treatment response assessment, also being of prognostic value. Subsequently following SIRT, patients are restaged with FDG-PET/CT. However, optimal timing of restaging following treatment is unknown (most commonly after 1 or 3 months, according to local institutional guidelines). More importantly, intrinsic resolution of FDG-PET/CT limits its utility in patients with small metastases, as image quality is worsened by high background noise, due to physiologic FDG uptake / metabolism in normal liver parenchyma. Additionally, FDG as radiopharmaceutical increases additional radiation burden to patients. This study will investigate the potential of metabolic MRI (7T MRI), non-invasively imaging metabolites using X-nuclei (e.g. 31P MRSI) and more importantly, the application of Deuterium Metabolic Imaging (DMI) with non-radioactive deuterated glucose, as a potential alternative over FDG-PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Referred for SIRT and deemed eligible by the multidisciplinary tumor board
* Size of at least one liver metastasis ≥ 1 cm on contrast enhanced CT / MRI (measurable according to RECIST 1.1) and 18FDG-avid metastatic liver disease (uptake > healthy liver uptake; measurable according to PERCIST)
* Written informed consent

Exclusion Criteria:

* Patients having FDG-negative disease (according to PERCIST)
* Patients with diabetes mellitus
* Patients having a general contra-indication for SIRT
* Patients with contra-indications for 7T MR scanning
* Patient unable to complete study scan (laying still for a long time)
* Patient unable or incapable to follow study proceedings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
To confirm feasibility of DMI for intrahepatic tumor detection. | 1 and 3 months after radioembolization, anatomical and molecular imaging is repeated.
  Image quality comparison between DMI and FDG-PET/CT, defined as technical performance (e.g. signal-to-noise and tumor-to-liver ratios) and intrahepatic lesion detection.

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Netherlands